CLINICAL TRIAL: NCT01460433
Title: A Compartmental Analysis of HIV Reservoirs and Immune Reconstitution (C)
Brief Title: Problems With Immune Recovery in the Gut Tissue
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0712M22449; P01AI074340 (NIH)
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV 1; Herpes Simplex Type 2; Treatment experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, lymphatic tissues and anogenital swabs.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Genital and rectal swabbing — Subjects swabs their genitals and rectum daily. The amount of HSV shed over the previous 24 hours is measured and the daily HSV shed rate is calculated.

SUMMARY:
The aim of this study is to find out if the process of HIV replication in the lymph tissue and gut tissue of people taking HIV drugs causes long-term damage to the ability of the gut to protect you from other infections and health problems.

ELIGIBILITY:
Inclusion Criteria:

HIV+ individuals

* Seropositive for HIV
* On ART for at least 12 months
* Seropositive for Herpes Simplex Type 2 and Cytomegalovirus
* Age ≥ 18 years
* Negative pregnancy test for eligible women of childbearing potential

HIV- individuals

* Seronegative for HIV
* Seropositive for Herpes Simplex Type 2 and Cytomegalovirus
* Age ≥ 18 years
* Negative pregnancy test for eligible women of childbearing potential

Exclusion Criteria:

* Taking daily suppressive therapy for Herpes Simplex Type 2
* Contraindication to surgical & endoscopic procedures (as judged by PI)
* Psychiatric or psychological illness that would make adherence to protocol procedures unlikely
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV+, antiretroviral-treated individuals who have been exposed to Herpes Simplex Type 2 and Cytomegalovirus and HIV- individuals who have been exposed to Herpes Simplex Type 2 and Cytomegalovirus.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2008-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Herpes Simplex Virus - Type 2 shed rate | 60 days

SECONDARY OUTCOMES:
Evidence of HIV replication in blood and lymphoid tissue | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Schacker, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States